CLINICAL TRIAL: NCT02521792
Title: A Phase 2, In-Home, Safety and Efficacy Evaluation of Episodic Administration of Open-Label Palovarotene in Subjects With Fibrodysplasia Ossificans Progressiva (FOP)
Brief Title: In-Home Evaluation of Episodic Administration of Palovarotene in Fibrodysplasia Ossificans Progressiva (FOP) Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Subjects were enrolled into a different Phase 2 study (PVO-1A-202, NCT02279095).
Sponsor: Clementia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PVO-1A-203
Record Dates: First submitted 2015-08-06; First posted 2015-08-13 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Fibrodysplasia Ossificans Progressiva
Keywords: Open-label study; Clinical trial Phase 2; Efficacy and safety; Heterotopic ossification; Fibrodysplasia Ossificans Progressiva; Flare-up; Palovarotene; Retinoic acid receptor agonist; Retinoic acid receptor gamma agonist; Clementia; Myositis Ossificans Progressiva; Munchmeyer's Disease; FOP
MeSH Terms: conditions — Myositis Ossificans; Ossification, Heterotopic | interventions — Palovarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Palovarotene (Experimental): The protocol is open only to the subjects who completed Clementia Study PVO-1A-202. Eligible subjects will receive a weight-based equivalent dose of palovarotene 10 mg once daily for 14 days, followed by 5 mg once daily for 28 days. Should treatment be extended beyond 6 weeks, a weight-based equivalent dose of 5 mg will be administered in 2-week increments.
  Interventions: Drug: Palovarotene

INTERVENTIONS:
Drug: Palovarotene — Palovarotene will be taken orally once daily at approximately the same time each day. Powder filled hard gelatin capsules may be opened and the contents added onto specific food.

SUMMARY:
Fibrodysplasia Ossificans Progressiva (FOP) is a rare, severely disabling disease characterized by painful, recurrent episodes of soft tissue swelling (flare-ups) that result in abnormal bone formation (heterotopic ossification or HO) in muscles, tendons, and ligaments. Flare-ups begin early in life and may occur spontaneously or after soft tissue trauma, vaccinations, or influenza infections. Recurrent flare-ups progressively restrict movement by locking joints leading to cumulative loss of function and disability. Mouse models of FOP have demonstrated the ability of retinoic acid receptor gamma (RARγ) agonists such as palovarotene to prevent HO following injury. This 36-month study will evaluate the long-term safety and efficacy of episodic treatment with palovarotene for flare-ups in FOP subjects who successfully complete two flare-up treatment periods (6 weeks duration) and two follow-up periods (6 weeks duration) in Study PVO-1A-202.

DETAILED DESCRIPTION:
The primary objective of this Phase 2, open-label, multicenter, single-arm, extension study is to investigate the safety and efficacy of episodic treatment with palovarotene in FOP subjects with flare-ups.

Secondary objectives are:

The effect of episodic treatment of flare-ups with palovarotene on range of motion (ROM) as assessed by the subject global assessment of movement.

* The effect of episodic treatment of flare-ups with palovarotene on ROM as assessed by the Cumulative Analogue Joint Involvement Scale for FOP (CAJIS) for subjects with video-conferencing capability.
* The effect of episodic treatment of flare-ups with palovarotene on the total burden of heterotopic ossification (HO) as assessed by low-dose whole body computerized tomography (WBCT), excluding the head; and whole body dual energy x-ray absorptiometry (DEXA).
* The effect of episodic treatment of flare-ups with palovarotene on physical function using age-appropriate forms of the FOP-Physical Function Questionnaire (FOP-PFQ).
* The effect of episodic treatment of flare-ups with palovarotene on physical and mental health using age appropriate forms of the Patient Reported Outcomes Measurement Information System (PROMIS) Global Health Scale.
* The effects of episodic treatment of flare-ups with palovarotene on pain and swelling associated with the flare-up using numeric rating scales (NRS) or the Faces Pain Scale-Revised (FPS-R) in subjects under 8 years of age.
* The use of assistive devices and adaptations for daily living by FOP subjects.

The follow-up portion of the study will consist of a Screening visit that will correspond to the last day (Study Day 84) of Study PVO-1A-202 and bi-annual assessments at Months 6, 12, 18, 24, 30, and 36.

Subjects experiencing a new, distinct flare-up during the 36-month follow-up will be evaluated and if eligible, receive palovarotene at the weight-adjusted equivalent of 10 mg for 14 days followed by 5 mg for at least 28 days. Any subject who received a lower dosing regimen due to tolerability issues during Study PVO-1A-202 will receive that tolerated dose.

For each flare-up there will be two periods:

1. A Screening period to occur within 7 days of the start of a new, distinct flare-up. The first dose of palovarotene will be taken within 10 days of the flare-up onset to allow for shipment of study medication to the subject's home.
2. A treatment period of at least 6 weeks duration. Subjects experiencing a new, distinct flare-up will be evaluated

ELIGIBILITY:
Inclusion Criteria:

For study enrollment

* Completed Study PVO-1A-202 having been treated with palovarotene (ie, 6 weeks on-treatment and 6-weeks follow-up) for two flare-ups.
* Written, signed, and dated informed consent or age-appropriate subject/parent assent (this must be performed according to local regulations).

For treatment with palovarotene for subsequent flare-ups

* Symptomatic onset of a new, distinct flare-up within 10 days of the first dose of study drug. Symptoms must be reported by the subject, be consistent with their previous flare-ups, and include a subject-reported onset date. The flare-up must be confirmed by the physician at screening via telephone contact and/or video-conferencing.
* Females of child-bearing potential (FOCBP) must have a negative blood (or urine) pregnancy test (with sensitivity of at least 50 mIU/mL) prior to administration of palovarotene. Male and FOCBP subjects must agree to remain abstinent during treatment and for 1 month after treatment or, if sexually active, to use two highly effective methods of birth control during and for 1 month after treatment. Additionally, sexually active FOCBP subjects must already be using two highly effective methods of birth control 1 month before treatment is to start. Specific risk of the use of retinoids during pregnancy, and the agreement to remain abstinent or use two highly effective methods of birth control will be clearly defined in the informed consent, and the subject or legally authorized representatives (eg, parents, caregivers, or legal guardians) must specifically sign this section.
* Subjects must be accessible for treatment with palovarotene and follow-up.

Exclusion Criteria:

For study enrollment

* Any reason that, in the opinion of the Investigator, would lead to the inability of the subject and/or family to comply with the protocol.

For treatment with palovarotene for subsequent flare-ups:

* Weight <20 kg.
* The flare-up is at a completely ankylosed joint.
* Intercurrent non-healed fracture at any location.
* If currently using vitamin A or beta carotene, multivitamins containing vitamin A or beta carotene, or herbal preparations, fish oil, and unable or unwilling to discontinue use of these products during palovarotene treatment.
* Exposure to synthetic oral retinoids in the past 30 days prior to screening (signature of the informed consent or age-appropriate subject assent).
* Concurrent treatment with tetracycline or any tetracycline derivatives due to the potential increased risk of pseudotumor cerebri
* History of allergy or hypersensitivity to retinoids or lactose.
* Female subjects who are breastfeeding.
* Subjects with uncontrolled cardiovascular, hepatic, pulmonary, gastrointestinal, endocrine, metabolic, ophthalmologic, immunologic, psychiatric, clinically significant abnormal laboratory findings, or other significant disease.
* Simultaneous participation in another interventional clinical research study within the past 4 weeks (except for Study PVO-1A-202).
* Subjects experiencing suicidal ideation (type 4 or 5) or any suicidal behavior within the past month prior to Screening as defined by the Columbia Suicide Severity Rating Scale.
* Any reason that, in the opinion of the Investigator, would lead to the inability of the subject and/or family to comply with the protocol.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2016-08-04 (Actual); Study Completion 2016-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (2):
- United States (2):
  - University of California San Francisco, Division of Endocrinology and Metabolism, San Francisco, California
  - University of Pennsylvania, Center for Research in FOP & Related Disorders, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Shimono K, Tung WE, Macolino C, Chi AH, Didizian JH, Mundy C, Chandraratna RA, Mishina Y, Enomoto-Iwamoto M, Pacifici M, Iwamoto M. Potent inhibition of heterotopic ossification by nuclear retinoic acid receptor-gamma agonists. Nat Med. 2011 Apr;17(4):454-60. doi: 10.1038/nm.2334. Epub 2011 Apr 3. PMID 21460849
- See also: Website for the International FOP Association — http://ifopa.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fibrodysplasia Ossificans Progressiva (FOP) subjects treated with palovarotene for 2 flare-ups in Study PVO-1A-202/Part A were enrolled. During enrolment, the dosage regimen for Study PVO-1A-202/Part B was optimized. Study PVO-1A-203 was terminated and participating subjects enrolled into Study PVO-1A-202/Part B to receive the modified regimen.
Pre-assignment Details: The screening visit for this study (PVO-1A-203) was the same day as the end of study visit for Study PVO-1A-202/Part A. Subjects experiencing an eligible flare-up received open-label palovarotene (treatment period of at least 6 weeks). Subjects were to be followed for 36 months with telephone/video-conferencing assessments performed every 6 months.
Groups:
- Palovarotene: Subjects experiencing an eligible flare-up received a weight-based equivalent dose of palovarotene 10 milligram (mg) orally once daily for 14 days, followed by 5 mg once daily for 28 days. If treatment was extended beyond 6 weeks (if deemed necessary by the Investigator), the palovarotene dose-equivalent of 5 mg was to be administered (in 2-week increments) until the flare-up resolved.
Period: Overall Study
Arm/Group | Palovarotene
Started | 6
Received Treatment | 4
Completed | 0
Not Completed | 6
Not completed — Study Terminated | 6

BASELINE CHARACTERISTICS:
Population: All enrolled subjects were included in the baseline analysis.
Groups:
- Palovarotene: Subjects experiencing an eligible flare-up received a weight-based equivalent dose of palovarotene 10 mg orally once daily for 14 days, followed by 5 mg once daily for 28 days. If treatment was extended beyond 6 weeks (if deemed necessary by the Investigator), the palovarotene dose-equivalent of 5 mg was to be administered (in 2-week increments) until the flare-up resolved.
Arm/Group | Palovarotene
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAEs)
Description: The primary endpoint was the safety of palovarotene as assessed by the incidence of TEAEs (including those known to be associated with retinoids) and serious adverse event (SAEs) monitored throughout the treatment period. TEAEs were adverse events reported during treatment with palovarotene or within 6 weeks after the end of treatment. Day 1 was the first day that study drug was administered for a flare-up. The number of subjects experiencing at least one TEAE or treatment-emergent SAE are presented.
Time Frame: Day 1 until 6 weeks after the end of treatment (an expected average treatment of 6 weeks). Assessed until data cut-off for study termination (maximum of 35 days).
Population: The safety population included all subjects who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Palovarotene
Number analyzed (Participants) | 4
Participants
  TEAE | 4
  Treatment-emergent SAE | 1

2. Secondary Outcome: Subject Global Assessment of Movement as Determined by a Subject Completed Questionnaire, or Proxy Completed Questionnaire in Subjects Under 8 Years of Age
Time Frame: Every 6 weeks while on study drug, at the end of treatment (should treatment be extended beyond 6 weeks), and 6 weeks after the end of treatment.
Population: The study was stopped prematurely and only 4 subjects received treatment. No summary statistics are available due to the limited data from the small number of evaluable subjects and individual subject data are not presented to protect the privacy of the individuals.
Arm/Group | Palovarotene
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline in Cumulative Analogue Joint Involvement Scale for FOP as Assessed by the Investigator Using Remote Video-conferencing
Time Frame: Baseline (flare-up screening), every 6 weeks while on study drug, at the end of treatment (should treatment be extended beyond 6 weeks), and 6 weeks after the end of treatment.
Population: as for outcome 2
Arm/Group | Palovarotene
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline in Extent of Heterotopic Ossification (HO) by Whole Body Low-dose Computerized Tomography (CT) Scan, Excluding the Head
Time Frame: Baseline (final visit for Study PVO-1A-202/Part A) and at end of study (36 months).
Population: as for outcome 2
Arm/Group | Palovarotene
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline in Extent of HO by Whole Body Dual Energy X-ray Absorptiometry (DEXA) Scan
Time Frame: Baseline (screening/enrollment visit) and at end of study (36 months).
Population: as for outcome 2
Arm/Group | Palovarotene
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in Pain and Swelling at the Flare-up Site Using Numeric Rating Scales, or Faces Pain Scale-Revised in Subjects Under 8 Years of Age
Time Frame: Baseline (flare-up screening), every 2 weeks while on study drug, at the end of treatment (should treatment be extended beyond 6 weeks), and 6 weeks after the end of treatment.
Population: as for outcome 2
Arm/Group | Palovarotene
Number analyzed (Participants) | 0

7. Secondary Outcome: Change From Baseline in Physical Function Using Age-appropriate Forms of the FOP-Physical Function Questionnaire
Time Frame: Baseline (flare-up screening), every 6 weeks while on study drug, at the end of treatment (should treatment be extended beyond 6 weeks), and 6 weeks after the end of treatment, and 6-month intervals for duration of study.
Population: as for outcome 2
Arm/Group | Palovarotene
Number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline in Physical and Mental Health Using Age-appropriate Forms of the Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Scale
Time Frame: Baseline (flare-up screening), every 6 weeks while on study drug, at the end of treatment (should treatment be extended beyond 6 weeks), 6 weeks after the end of treatment, and 6-month intervals for duration of study.
Population: as for outcome 2
Arm/Group | Palovarotene
Number analyzed (Participants) | 0

9. Secondary Outcome: Duration of Active, Symptomatic Flare-up as Assessed by the Subject and the Investigator
Time Frame: Baseline (flare-up screening), after 6 weeks on study drug, and every 2 weeks after Week 6 until flare-up resolution.
Population: as for outcome 2
Arm/Group | Palovarotene
Number analyzed (Participants) | 0

10. Secondary Outcome: Change From Baseline in the Use of Assistive Devices and Adaptations for Daily Living by FOP Subjects
Time Frame: Baseline (flare-up screening), 6 weeks after the end of treatment, and 6-month intervals for duration of study.
Population: as for outcome 2
Arm/Group | Palovarotene
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: TEAEs were to be collected from Day 1 until 6 weeks after the end of treatment (an expected average treatment of 6 weeks). Assessed until data cut-off for study termination (maximum of 35 days).
Description: The safety population included all subjects who received at least one dose of study drug.
Groups:
- Palovarotene: Eligible subjects received a weight-based equivalent dose of palovarotene 10 mg orally once daily for 14 days, followed by 5 mg once daily for 28 days during flare-ups. If treatment was extended beyond 6 weeks (if deemed necessary by the Investigator), a weight-based equivalent dose of 5 mg was to be administered in 2-week increments.
Arm/Group | Palovarotene
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palovarotene (N=4)
Myoclonus (Nervous system disorders) | 1 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palovarotene (N=4)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3)
Lip dry (Gastrointestinal disorders) | 2 (2)
Dry eye (Eye disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was stopped prematurely and due to the small number of evaluable subjects, there was insufficient data to conduct any efficacy analyses. Consequently, no summary statistics are available for any of the secondary outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes